CLINICAL TRIAL: NCT00639366
Title: Prospective Randomised Clinical Trial Testing the Role of Prophylactic Cranial Radiotherapy in Patients Treated With Trastuzumab (Herceptin®) for Metastatic Breast Cancer
Brief Title: Radiation Therapy to the Head in Preventing Brain Metastases in Women Receiving Trastuzumab and Chemotherapy for Metastatic or Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anglo Celtic Cooperative Oncology Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: ACCOG-HER-PCI; CDR0000588868 (Registry Identifier: PDQ (Physician Data Query)); ISRCTN64624715; EU-20822
Record Dates: First submitted 2008-03-19; First posted 2008-03-20 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2008-12

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Drug Therapy; Radiotherapy

INTERVENTIONS:
Biological: trastuzumab
Drug: chemotherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. It is not yet known whether radiation therapy directed at the head is effective in preventing brain metastases in patients with advanced cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy to the head to see how well it works in preventing brain metastases in women receiving trastuzumab and chemotherapy for metastatic or locally advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test if prophylactic cranial radiotherapy delivering 30 Gy in 10 fractions will significantly reduce (from 35% to 21% at 2 years) the incidence of symptomatic brain metastases in patients treated with trastuzumab (Herceptin®) for metastatic breast cancer.

OUTLINE: This is a multicenter study. Patients are stratified by center, type of systemic therapy (trastuzumab [Herceptin®] monotherapy vs combination with chemotherapy), hormone receptor status, and presence of lung metastases (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive taxane/trastuzumab therapy for 6 weeks. While continuing taxane/trastuzumab therapy, patients then undergo 10 fractions of concurrent prophylactic cranial radiotherapy in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive taxane/trastuzumab therapy without concurrent prophylactic cranial radiotherapy.

All patients undergo quality of life assessments every 8 weeks for 9 months.

After completion of study treatment, patients are followed periodically for at least 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven breast carcinoma

  * Metastatic or locally advanced disease
* Must demonstrate HER2 3+ positivity on IHC or 2+ over-expression and FISH test demonstrating C-erB2 gene amplification
* No known or suspected brain metastases or CNS disease, as defined by the presence of any of the following key symptoms:

  * Headache
  * Nausea and/or vomiting
  * Clinical signs of raised intracranial pressure
  * Seizures
  * Focal symptoms
  * Cognitive dysfunction
  * Affective disorder
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal status not specified
* ECOG performance status 0 or 1
* Patients must a-priori be suitable for trastuzumab (Herceptin®) +/- chemotherapy in terms of bone marrow, hepatic, and renal function
* No prior history of cerebrovascular disease or neurological disorder including seizures

PRIOR CONCURRENT THERAPY:

* No prior cranial radiotherapy
* No prior neurosurgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2007-02; Primary Completion 2010-02 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Incidence of symptomatic brain metastases

SECONDARY OUTCOMES:
Survival
Cerebral toxicity and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Canney, MD, Principal Investigator — University of Glasgow
Locations (19):
- United Kingdom (19):
  - Basildon University Hospital, Basildon, England
  - Ipswich Hospital, Ipswich, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Aintree University Hospital, Liverpool, England
  - Barts and the London School of Medicine, London, England
  - Christie Hospital, Manchester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Great Western Hospital, Swindon, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Cancer Care Centre at York Hospital, York, England
  - Dumfries & Galloway Royal Infirmary, Dumfries, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Falkirk and District Royal Infirmary, Falkirk, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Crosshouse Hospital, Kilmarnock, Scotland
  - Wishaw General Hospital, Wishaw, Scotland